CLINICAL TRIAL: NCT06989307
Title: COVID-19 Serologies Among Healthcare Workers at CHSD (SERO2)
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0011_SMIT
Record Dates: First submitted 2025-05-22; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: COVID-19; COVID-19 Serological Testing; COVID-19 Vaccines; Health Personnel; Antibodies, Viral; Seroepidemiologic Studies
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looks at how many healthcare workers at CHSD hospital developed antibodies against COVID-19 after the second and third waves of the pandemic and after receiving a vaccine. It aims to better understand who might still be at risk of infection, how long immunity lasts after getting COVID or the vaccine, and how reliable previous antibody tests were. Blood samples will be collected from volunteer hospital staff during a one-month period to measure their antibody levels and compare them to earlier results.

ELIGIBILITY:
Inclusion Criteria:

- Volunteers from the hospital staff who have signed a new informed consent form

Exclusion Criteria:

* Refusal to participate (no signed consent form)
* Staff unavailable during the blood sampling period
* Participation only in the first seroprevalence survey without consent for the second

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study participants will be selected from the staff of the CHSD hospital. The target population includes all hospital personnel, regardless of role or department, who volunteer to participate and provide informed consent for the serological survey.
Sampling Method: Non-Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 antibody prevalence (seroprevalence) among healthcare workers at CHSD | 1 month (during the serological testing period)

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France